CLINICAL TRIAL: NCT01385150
Title: Analysis of Serum 2-Hydroxyglutarate (2HG) Levels, IDH Mutations and Clinical Outcome in Acute Myeloid Leukemia (AML)
Brief Title: Biomarkers in Blood Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000702952; ECOG-E1900T8
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute | interventions — Chromatography, Liquid; Mass Spectrometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: mutation analysis
Genetic: protein analysis
Other: laboratory biomarker analysis
Other: liquid chromatography
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors identify and lean more about biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in blood samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if serum 2-hydroxyglutarate (2HG) is only detected in acute myeloid leukemia (AML) patients with isocitrate dehydrogenase (IDH) mutations.

Secondary

* To determine if the level of serum 2HG impacts leukemia-free survival (LFS).
* To determine if the level of serum 2HG impacts overall survival (OS).
* To determine if serum 2HG is undetectable at the time of documented clinical remission (CR) in IDH-mutated patients.

OUTLINE: Archived serum samples are analyzed for 2-hydroxyglutarate expression by reverse-phase liquid chromatography coupled to mass spectrometry. Results are then compared with presence or absence of an IDH mutation, patients' clinical outcome, as well as age, sex, white blood cell count at diagnosis, platelet count, bone marrow blast percentage at diagnosis, circulating (serum) percentage at diagnosis, cytogenetic risk group, presence of FLT3, NPMN1, and/or TET2 mutations, specific IDH mutation, and randomization treatment group allocation.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute myeloid leukemia (AML)

  * Newly diagnosed with AML
  * Serum samples from patients enrolled on the ECOG-1900 clinical trial between 2002 and 2008
  * Patients with or without isocitrate dehydrogenase (IDH) mutations

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Received 2 different doses of standard induction chemotherapy on ECOG-1900

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Samples from patients enrolled on E1900 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2012-01-03 (Actual); Primary Completion 2012-02-03 (Actual); Study Completion 2012-02-03 (Actual)

PRIMARY OUTCOMES:
Absence of serum 2HG in all samples without an IDH mutation | 1 day

SECONDARY OUTCOMES:
Relationship between 2HG level and survival outcomes | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine